CLINICAL TRIAL: NCT05353907
Title: Dual-Energy Computed Tomography for Improving Imaging Assessment of Multiple Myeloma
Acronym: DECIMA
Status: Not yet recruiting | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 274302
Record Dates: First submitted 2022-02-04; First posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Myeloma
MeSH Terms: conditions — Neoplasms, Plasma Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Whole Body MRI — Once recruited, the participant will undergo a WB-MRI scan as part of their usual standard-of-care. As part of the research study, the participant will be consented to undertake an additional WB-DECT research scan at a time of their choosing (on the same day as the MRI scan, or on another day, if preferred)
  Other Names: Whole Body Dual Energy CT

SUMMARY:
Up to 30% of patients with newly diagnosed/suspected myeloma cannot undergo or do not tolerate whole body MRI (WB-MRI). A number of factors may be contributory. First, WB-MRI protocols can take in excess of 1 hour. Patients must remain still within a narrow bore scanner with multiple MRI coils that can be claustrophobic. Second, there is significant acoustic noise that can be heard despite the use of ear protection. Third, 80% of patients will experience bone pain or fracture at some point during their illness, affecting their comfort within the scanner. Fourth, patients also have higher anxiety. One review reported up to 30% of patients experienced considerable apprehension and up to 10% severe psychological distress when undergoing MRI. Finally, myeloma is predominantly an illness of the elderly and co-morbid conditions decrease patients' ability to tolerate a long scan. When WB-MRI cannot be performed, NICE recommend whole-body computed tomography (WB-CT), which the investigators know offers decreased diagnostic performance in terms of marrow assessment and focal lesion detection. The investigators believe that using a novel CT technique - dual-energy CT (DECT) - may offer better diagnostic performance over standard WB-CT in myeloma patients.

What the investigators seek to do in this study is to evaluate the sensitivity and specificity of DECT in a cohort of untreated patients; and compare the performance of DECT to simulated standard CT (data simulated from the DECT) and also to WB-MRI (reference standard alongside bone marrow biopsy results. The investigators will assess both subjective visual analysis of DECT images as well as CT quantitative values for the bone marrow.

Secondary objectives include assessment of patient experience across both imaging tests and assessment of intra & inter observer variability in subjective visual analysis

ELIGIBILITY:
Inclusion Criteria:

* Adults with suspected or newly diagnosed myeloma

Exclusion Criteria:

* No previous treatment for myeloma
* No concurrent cancer elsewhere
* No contraindications to CT or MRI scans
* Routine, standard of care cut-off for minimum renal function (eGFR > 40 ml/min/1.73 m2) in order to receive IV gadolinium-based contrast media.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with suspected or newly diagnosed myeloma
Sampling Method: Non-Probability Sample
Enrollment: 78 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of WB-DECT | Baseline (both scans acquired at the same time point)
  Sensitivity and specificity of whole body dual-energy CT (WB-DECT) to detect focal lesions and marrow infiltration compared to WB-MRI (gold standard) and WB-CT.

SECONDARY OUTCOMES:
Qualitatively measure patient experience of WB-DECT compared to WB-MRI . | Baseline (both scans acquired at the same time point)
  Pre and post scan questionnaire administered for both WB-MRI and WB-DECT. Thematic analysis will be used.
Intra & inter observer variability in subjective visual analysis and quantitative analysis of WB-DECT | Baseline (both scans acquired at the same time point)
  Measured by Kappa statistic.

CONTACTS AND LOCATIONS:
Overall Officials: Vicky Goh, Principal Investigator — King's College London